CLINICAL TRIAL: NCT02540135
Title: Fluorescein vs. Intraoperative MRI in the Resection of Malignant High Grade Glioma
Brief Title: Fluorescein vs. iMRI in Resection of Malignant High Grade Glioma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The investigators decided not to move forward with this study at this time.
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 15-1313
Record Dates: First submitted 2015-09-01; First posted 2015-09-03 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: High Grade Malignant Neoplasm; Glioblastoma Multiforme; Anaplastic Astrocytoma
Keywords: high grade glioma; glioblastoma multiforme; anaplastic astrocytoma; flourescein; flourescence-guided surgery; intraoperative MRI; iMRI
MeSH Terms: conditions — Glioblastoma; Astrocytoma; Glioma | interventions — Fluorescein

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Experimental): Flourescein plus intraoperative MRI
  Interventions: Other: fluorescein; Other: intraoperative MRI
- Arm B (Active Comparator): intraoperative MRI alone
  Interventions: Other: intraoperative MRI

INTERVENTIONS:
Other: fluorescein — fluorescein and conventional neuro-navigation
  Arms: Arm A
Other: intraoperative MRI — conventional neuro-navigation and iMRI
  Other Names: iMRI

SUMMARY:
This study plans to learn more about if fluorescein with intraoperative Magnetic Resonance Imaging (MRI) is as good as intraoperative MRI (iMRI) alone in detecting the presence of tumor tissue during surgery.

Both fluorescein and intraoperative MRI have been studied and routinely used to aid the neurosurgeon in distinguishing normal brain from tumor, helping the neurosurgeon to safely resect more tumor tissue during surgery.

This study will enroll patients with malignant high grade glioma who are going to have a surgery to remove their brain tumor.

For half of the patients, fluorescein and intraoperative MRI will be used together during surgery. For half of the patients, only intraoperative MRI will be used during surgery. iMRI is used as final verification of complete, safe resection in both arms.

DETAILED DESCRIPTION:
Extent of surgical resection of malignant high grade glioma has been established as one of the most important predictors of overall survival and six-month progression free survival. Unfortunately, it is often difficult in surgery to distinguish between tumor and normal brain. Various technologies have been developed to help the surgeon more readily safely increase extent of resection in order to achieve an improved survival after glioblastoma resection. Fluorescein has been used at some institutions for a number of years to improve visualization of high-grade gliomas enabling their better resection. Intraoperative MRI has also been developed with similar intent, allowing the patient to be imaged intraoperatively to determine extent of resection and any need for further resection prior to leaving the operating room. While there is some evidence these technologies improve extent of resection in comparison to historical controls, they have never been tested against each other in any prospective fashion.

Intraoperative MRI has significant cost and significantly increases operative time. Fluorescein is a very inexpensive injectable agent and, if as good at achieving gross total resection as intraoperative MRI, would offer patients similar surgical outcomes with less anesthetic time and cost than intraoperative MRI. This study aims to investigate the value of fluorescein or intraoperative MRI in malignant glioma patients' extent of tumor resection in a prospectively randomized manner.

ELIGIBILITY:
Inclusion Criteria:

* Presents with presumed or pathologically proven enhancing primary or secondary high grade glioma for surgical resection
* Eligible for gross total resection of enhancing component of tumor
* Karnofsy performance status >/= 70%

Exclusion Criteria:

* Presence of multi-focal disease
* Disease that crosses the mid-line
* History of adverse reaction to flourescein
* Known ongoing pregnancy
* Inability to grant consent
* Contraindication to perform iMRI
* Contraindication to flourescein

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03-01 (Estimated); Primary Completion 2018-07-18 (Actual); Study Completion 2018-07-18 (Actual)

PRIMARY OUTCOMES:
Extent of resection | 36 hours
  This outcome will utilize tumor volumetry of residual enhancing tumor after resection.

SECONDARY OUTCOMES:
Surgical time difference | 36 hours
  This outcome will evaluate the difference in length of surgery time between each arm.

CONTACTS AND LOCATIONS:
Overall Officials: David R Ormond, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States